CLINICAL TRIAL: NCT05465902
Title: Safety and Immunogenicity of Recombinant COVID-19 Variant Vaccine (Sf9 Cell) as a Booster Following Primary Vaccination of Either Inactivated or mRNA or Viral Vector COVID-19 Vaccines
Brief Title: Safety and Immunogenicity of Recombinant COVID-19 Variant Vaccine (Sf9 Cell) as a Booster
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trials not conducted
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT149
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Inactivated COVID-19 vaccines cohort group 1 (Experimental): Participants who received 2 doses of Inactivated COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment, N=100 Intervention: Recombinant COVID-19 variant Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 variant Vaccine (Sf9 Cell)
- Inactivated COVID-19 vaccines cohort group 2 (Active Comparator): Participants who received 2 doses of Inactivated COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment, N=100 Intervention: COVID-19 Vaccine (Vero Cell), Inactivated
  Interventions: Biological: COVID-19 Vaccine (Vero Cell), Inactivated
- mRNA COVID-19 vaccines cohort group 1 (Experimental): Participants who received 2 doses of mRNA COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=100 Intervention: Recombinant COVID-19 variant Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 variant Vaccine (Sf9 Cell)
- mRNA COVID-19 vaccines cohort group 2 (Active Comparator): Participants who received 2 doses of mRNA COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=100 Intervention: mRNA COVID-19 vaccine (Moderna)
  Interventions: Biological: mRNA COVID-19 vaccine (Moderna)
- Viral Vector COVID-19 vaccines cohort group 1 (Experimental): Participants who received 2 doses of Viral Vector COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=100 Intervention: Recombinant COVID-19 variant Vaccine (Sf9 Cell)
  Interventions: Biological: Recombinant COVID-19 variant Vaccine (Sf9 Cell)
- Viral Vector COVID-19 vaccines cohort group 2 (Active Comparator): Participants who received 2 doses of Viral Vector COVID-19 vaccines with the second dose at least 6 months (≥180 days) prior to enrolment. N=100 Intervention: Viral Vector COVID-19 vaccine (AstraZeneca)
  Interventions: Biological: Viral Vector COVID-19 vaccine (AstraZeneca)

INTERVENTIONS:
Biological: Recombinant COVID-19 variant Vaccine (Sf9 Cell) — 1dose, Intramuscular Injection
  Arms: Inactivated COVID-19 vaccines cohort group 1; Viral Vector COVID-19 vaccines cohort group 1; mRNA COVID-19 vaccines cohort group 1
Biological: COVID-19 Vaccine (Vero Cell), Inactivated — 1dose, Intramuscular Injection
  Arms: Inactivated COVID-19 vaccines cohort group 2
Biological: mRNA COVID-19 vaccine (Moderna) — 1dose, Intramuscular Injection
  Arms: mRNA COVID-19 vaccines cohort group 2
Biological: Viral Vector COVID-19 vaccine (AstraZeneca) — 1dose, Intramuscular Injection
  Arms: Viral Vector COVID-19 vaccines cohort group 2

SUMMARY:
This is a randomized, phase Ⅱ, single-blind, randomized, parallel-group controlled clinical trial.

The study plans to enroll subjects who have completed homologous primary vaccination with either inactivated or mRNA or Viral Vector COVID-19 vaccines (one or two doses) and have not been infected with COVID-19. All subjects will be evaluated for safety and immunogenicity after a single dose booster immunization with Recombinant COVID-19 variant Vaccine (Sf9 Cell) or inactivated COVID-19 vaccine (Vero cell) or mRNA vaccine or Viral Vector vaccine.

DETAILED DESCRIPTION:
This is a randomized, phase Ⅱ, single-blind, randomized, parallel-group controlled clinical trial.

The study plans to enroll subjects who have completed homologous primary vaccination with either inactivated or mRNA or Viral Vector COVID-19 vaccines (one or two doses) and have not been infected with COVID-19. All subjects will be evaluated for safety and immunogenicity after a single dose booster immunization with Recombinant COVID-19 variant Vaccine (Sf9 Cell) or inactivated COVID-19 vaccine (Vero cell) or mRNA vaccine or Viral Vector vaccine. The study plans to enroll about 600 subjects aged 18 years and above (subjects aged ≥ 60 years account for approximately 10%) that would be divided into three cohorts according to different primary vaccination: Inactivated COVID-19 vaccines cohort, mRNA COVID-19 vaccines cohort and Viral Vector COVID-19 vaccines cohort, with approximately 200 cases in each cohort. The subjects will be randomized to the Recombinant COVID-19 variant Vaccine (Sf9 Cell) group (test group) or the inactivated COVID-19 vaccine (Vero cell) group or mRNA vaccine or Viral Vector vaccine (control group) in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily sign the ICF approved by the Ethics Committee and agree to participate in the study before any study procedure.
* 2. Healthy males or females able to provide legal identification, aged 18 years and above at the time of signing ICF.
* 3. Subjects who have completed homologous primary vaccination with either Inactivated or mRNA or Viral Vector COVID-19 vaccines (full approval, CMA or EUA) and have the last dose administered 6 months ago or earlier from the date of signing the ICF for the study. Those who have received combined immunization with two doses of vaccines should be excluded.
* 4. Able to communicate well with the investigator, and able to understand and comply with the requirements of this clinical trial.
* 5. Males with female sexual partners or females of childbearing potential voluntarily take effective contraceptive methods from signing ICF to 3 months after the vaccination, including sexual abstinence or effective contraceptive measures (e.g., intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, intrauterine device (IUD), condoms (male), diaphragm, and cervical cap).
* 6. Axillary temperature <37.3℃.

Exclusion Criteria:

* 1. Positive SARS-CoV-2 RT-PCR at screening.
* 2. Prior medical history of Serve Acute Respiratory Syndromes (SARS), Middle East Respiratory Syndrome (MERS) and other human coronavirus infections or diseases.
* 3. Prior history or family history of convulsion, epilepsy, encephalopathy and psychosis.
* 4. Fear of needles.
* 5. Pregnant or lactating females or those who plan to become pregnant or donate eggs during study period.
* 6. Prior history of allergic reaction or anaphylaxis to any vaccine or its excipients, e.g., hypersensitivity, urticaria, serious eczema, dyspnea, laryngeal edema, and angioedema etc..
* 7. Prior use of any vaccine within 28 days before receiving this investigational vaccine or planning to use any vaccine other than this investigational vaccine during the study period.
* 8. Participation in studies of any other interventional device or drug within 28 days before the screening, or current treatment with other investigational drug(s) or within 5 half-lives after taking the last dose of the study drug.
* 9. Hereditary hemorrhagic tendency or coagulation dysfunction (e.g., clotting factors deficiency, coagulation disorders or platelet disorders), or a history of severe bleeding, or a history of massive bleeding after intramuscular injection or venipuncture, or a history of ecchymosis.
* 10. Known medical history or diagnosis confirming that subjects have diseases affecting immune system function, including cancer, congenital or acquired immunodeficiency (e.g., infection with Human Immunodeficiency Virus (HIV)), or uncontrolled autoimmune disease.
* 11. Serious or uncontrolled respiratory system disorders, cardiovascular disorders, nervous system disorders, blood and lymphatic system disorders, liver and kidney disorders, metabolism and skeletal disorders, etc. influencing study results evaluation at the investigator's discretion.
* 12. Asplenia or functional asplenia.
* 13. Long-term use (continuous use for ≥14 days) of immunosuppressants or other immunomodulators (e.g., glucocorticoids: prednisone or equivalents) within 6 months prior to administration of this investigational vaccine, except for topical medications (e.g., ointments, eye drops, inhalants or nasal sprays). And the topical medications should not exceed the recommended dose in the labels or induce any signs of systemic exposure.
* 14. Having received immunoglobulins and/or blood products within 3 months prior to administration of this investigational vaccine.
* 15. History of tuberculosis treatment or currently on antikoch's treatment for tuberculosis, whether pulmonary or extrapulmonary.
* 16. Suspected or known alcohol dependency or drug abuse, which may affect safety evaluation or subject's compliance at the investigator's discretion.
* 17. Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits.
* 18. An employee of the study site, Sponsor and contract research organization (CRO) taking part in the study.
* 19. Other conditions unsuitable for this study at the investigator's discretion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) | Day 0-28 post-boost dose
GMT and SCR of specific neutralizing antibody (virus or pseudovirus) against SARS-CoV-2 | Day 14 post-boost dose

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Day 0-7 post-boost dose
Incidence of AEs | Day 0-28 post-boost dose
Incidence of serious adverse events (SAEs) | Day 0 through 6 months post-boost dose
GMT and SCR of specific neutralizing antibody (virus or pseudovirus) against SARS-CoV-2 | Day 28, month 3 and month 6 post-boost dose
GMI of specific neutralizing antibody (virus or pseudovirus) against SARS-CoV-2 | Day 14, Day 28, month 3 and month 6 post-boost dose
GMT, GMI and SCR of IgG antibodies against Vac2107 of SARS-CoV-2 | Day 14, Day 28, month 3 and month 6 post-boost dose

OTHER OUTCOMES:
GMT, GMI, and SCR of specific neutralizing antibody (virus or pseudovirus) against SARS-CoV-2 endemic variants | Day 14, Day 28, month 3 and month 6 post-boost dose

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica de Enfermedades Crónicas y de Procedimientos Especiales, S.C., Morelia, Michoacán, Mexico